CLINICAL TRIAL: NCT02327975
Title: Effects of a Training Program of Physical Exercise Administered Through Mobile Application in Elderly
Brief Title: Prescription of Physical Exercise Through Mobile Application in Elderly
Acronym: PEME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Balearic Islands (Other)
Responsible Party: Principal Investigator, Josep1, Professor, University of the Balearic Islands
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: I+D
Record Dates: First submitted 2014-12-20; First posted 2014-12-31 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Motor Activity; Aerobic Exercise; Mobile Applications; Aged; Prescriptions; Cell Phones; Resistance Training; Muscle Strenght
MeSH Terms: conditions — Motor Activity | interventions — Sensitivity Training Groups; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Training group (Experimental): Participants in this group received twice-weekly non-consecutive sessions of physical exercise for 10 weeks. Each session lasted approximately 60-70 minutes. Exercise program consisted of strength training and aerobic exercise. Each session began with a warm low intensity (10 min), then the main part of the session (25 min) and aerobic training and recovery period (25-35 min) was performed. The equipment used during the procedure was the Thera-Band elastic band.
  Interventions: Other: Training group
- Mobile group (Experimental): Intervention content was the same in both intervention arms; only the delivery mode differed. Participants in this group received two podcast (digital multimedia file available for download in a media player) per week for 10 weeks of the intervention, each podcast lasted about 5 min. Participants in this group received a weekly message with the aim of fostering motivation toward physical activity. Subjects in this group performed two sessions per week on non-consecutive days, the days could be chosen by the participants themselves.
  Interventions: Other: Mobile group
- Control group (Other): No received intervention.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Training group — The main part of the session included a whole-body strength training, which incorporated chest press, shoulder press, lateral pull-down, seated row, shoulder flexion, chest pulley, hammer curl, biceps curl, triceps curl, triceps pushdown, leg extension, leg curl, lunge, squat, abdominal crunch. To control and equate the intensity between the TG and MG, a method based on the combined use of the prescribed number of repetitions and the OMNI Resistance Scale for the active muscles was used. Previous studies have described the method used for controlling exercise intensity (Colado et al., 2012; Colado et al., 2014).
  During 1-3 weeks subjects performed 25 min of exercise at 60% maximum heart rate (HRmax), during weeks 4-6 subjects performed 30 min of exercise at 70% HRmax and during weeks 7-10 subjects performed 35 min of exercise at 80% HRmax.
  Arms: Training group
Other: Mobile group — The subjects in this group received the same intervention that trainning group but through a mobile application (whatsapp).
  Arms: Mobile group
Other: Control group — No received intervention.
  Arms: Control group

SUMMARY:
Physical inactivity is a health problem that affects people worldwide and has been identified as the fourth largest risk factor for overall mortality (contributing to 6% of deaths globally). Many researchers have tried to increase physical activity (PA) levels through traditional methods without much success. Thus, many researchers are turning to mobile technology as an emerging method for changing health behaviours.The study consists of a physical activity intervention through a mobile application in elderly. The study is a 3x2 model, in which the sample is distributed in three study groups (over 53 years) and were evaluated at 10 weeks from baseline.

DETAILED DESCRIPTION:
Objectives of the study:

* Evaluate effectiveness of a physical exercise program for 10 weeks to improve fitness, cardiovascular, anthropometric and body composition parameters in people over 53 years.
* Examine effects of exercise intervention delivered through a mobile application (WhatsApp) on fitness, cardiovascular risk factors, anthropometric and body composition in people over 53 years.

Hypotheses of the study:

* An intervention of exercise administered via mobile application (WhatsApp) is effective in reducing cardiovascular risk factors in people over 53 years.
* An intervention of exercise administered via mobile application (WhatsApp) is effective to increase physical fitness in people over 53 years.
* An intervention of exercise administered via mobile application (WhatsApp) is effective in reducing BMI, percent body fat; and in increasing the percentage of muscle mass in people over 53 years.
* 10-weeks face-to-face intervention of physical exercise obtains greater improvements in fitness parameters than an intervention delivered via mobile application in people over 53 years.
* 10-weeks face-to-face intervention of physical exercise obtains greater improvements in anthropometric and body composition than an intervention delivered via mobile application in people over 53 years.

ELIGIBILITY:
Inclusion Criteria:

* Have own mobile phone and Internet
* Be clinically stable
* Be able to perform physical activity
* Be able to understand and complete the informed consent
* Ability to cope assessment tests

Exclusion Criteria:

* Unable to perform physical activity
* Have an acute or chronic disease
* Have medical conditions or other physical problem that needs special attention (history of fracture of any upper or lower limb, dementia, psychological problems, neuromuscular disease, history of myocardial infarction, osteoporosis, cancer, diabetes).

Min Age: 53 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Maximum hand grip strength (dynamometry) | Change from Baseline in Maximum hand grip strength (dynamometry) at 10 weeks
  The manual pressure force was measured with a digital force gauge (TKK 5001 Grip-A; Takey, Tokyo, Japan) and the results are recorded in kilograms
Change from Baseline in Aerobic capacity | Change from Baseline in Aerobic capacity at 10 weeks
  Aerobic capacity was measured using 2-Minute Step Test.
Change from Baseline in Static Balance | Change from Baseline in Static Balance at 10 weeks
  Static balance measurement was conducted using the Flamingo test (Committee of Experts on Sport Research, 1988).
Change from Baseline in Waist circumference | Change from Baseline in Waist circumference at 10 weeks
Change from Baseline in Body fat | Change from Baseline in Body fat at 10 weeks
  Body fat was measured using Bioimpedance scale (Tanita Body Fat Monitor Scale plus, Model BF-556) is used
Change from Baseline in Muscle mass | Change from Baseline in Muscle mass at 10 weeks
  Muscle mass was measured using Bioimpedance scale (Tanita Body Fat Monitor Scale plus, Model BF-556) is used

SECONDARY OUTCOMES:
Change from Baseline in Physical activity levels | Change from Baseline in Physical activity levels at 10 weeks
  To measure levels of physical activity of the participants used the International Physical Activity Questionnaire (IPAQ) (Craig et al., 2003)
Change from Baseline in Height | Change from Baseline in Height at 10 weeks
  The height was measured as close to the millimeter using the mobile rod (Seca 217).
Change from Baseline in Weight | Change from Baseline in Weight at 10 weeks
  The weight was measured using bioelectrical impedance scales (Tanita Body Fat Monitor Scale plus, Model BF-556).
Change from Baseline in Systolic Blood Pressure | Change from Baseline in Systolic Blood Pressure at 10 weeks
  The Systolic Blood Pressure was measured using Omron Elite 7300W (Omron Healthcare Inc, Bannockburn, IL, USA)
Change from Baseline in Dyastolic Blood Pressure | Change from Baseline in Dyastolic Blood Pressure at 10 weeks
  The Dyastolic Blood Pressure was measured using Omron Elite 7300W (Omron Healthcare Inc, Bannockburn, IL, USA)

CONTACTS AND LOCATIONS:
Overall Officials: Josep Vidal Conti, Principal Investigator — University of Balearic Islands
Locations (1):
- Josep Vidal Conti, Majorca, Balearic Islands, Spain

REFERENCES:
- [Derived] Muntaner-Mas A, Vidal-Conti J, Borras PA, Ortega FB, Palou P. Effects of a Whatsapp-delivered physical activity intervention to enhance health-related physical fitness components and cardiovascular disease risk factors in older adults. J Sports Med Phys Fitness. 2017 Jan-Feb;57(1-2):90-102. doi: 10.23736/S0022-4707.16.05918-1. Epub 2015 Sep 11. PMID 26364690